CLINICAL TRIAL: NCT06974487
Title: A Randomized, Double-Blind, Crossover Phase I Clinical Study to Evaluate the Safety, Tolerability, PK and PD Profiles of a Single Dose of GZR102 Injection Versus GZR4 Injection and GZR18 Injection Given Separately in Chinese Adult Overweight Subjects
Brief Title: A Phase I Study to Evaluate the PK and PD Profiles of GZR102 Injection Versus GZR4 Injection and GZR18 Injection Given Separately in Chinese Adult Overweight Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GZR102-T2D-101
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GZR102 injection (Experimental): Participants will get a single dose of GZR102 injection （fixed-ratio combination of GZR4 and GZR18）.
  Interventions: Drug: GZR102 injection
- GZR4 injection (Active Comparator): Participants will get a single dose of GZR4 injection
  Interventions: Drug: GZR18 injection
- GZR18 injection (Active Comparator): Participants will get a single dose of GZR18 injection
  Interventions: Drug: GZR4 injection

INTERVENTIONS:
Drug: GZR102 injection — Participants will get a single dose of GZR102 injection （fixed-ratio combination of GZR4 and GZR18）.
  Arms: GZR102 injection
Drug: GZR4 injection — Participants will get a single dose of GZR4 injection
  Arms: GZR18 injection
Drug: GZR18 injection — Participants will get a single dose of GZR18 injection
  Arms: GZR4 injection

SUMMARY:
This trial is a randomized, double-blind, three-period crossover Phase I Clinical Study conducted in Chinese adult overweight subjects to evaluate the safety, tolerability, PK and PD profiles of a single dose of GZR102 injection versus GZR4 injection and GZR18 injection given separately.

Subjects undergo a screening phase of up to 3 weeks (D-21 to D-3). Eligible subjects are randomized in a 1:1:1:1:1:1 ratio into six dosing sequences, receiving single doses of GZR102 injection, GZR4 injection, and GZR18 injection across 3 cycles. A washout period of at least 1 week separates each cycle.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects sign the Informed Consent Form (ICF) before the study, fully understand the contents, process and possible adverse reactions of the study, and be able to follow the contraindications and restrictions specified in this protocol.

  2. Subjects (male or female) age 18-60 years old (inclusive) at the time of signing ICF.

  3. Body weight ≥ 60 kg, body mass index (BMI) ≥ 24 kg/m2 and < 28 kg/m2 at screening.

  4. No birth plan from the signing of ICF to 8 weeks after the last dose, willingness to use effective methods of contraception, and no plan for sperm donation. Females of childbearing potential must not be lactating and must have negative results of blood pregnancy tests at screening and predose.

Exclusion Criteria:

* 1. History of drug abuse prior to screening; or positive results for drug abuse at screening.

  2. History of alcohol abuse defined as an average alcohol intake of more than 14 units per week (1 standard unit = 360 mL of beer or 150 mL of 12% wine or 45 mL of 40% spirits) within 6 months prior to screening.

  3. Subjects who smoked > 5 cigarettes/day within 3 months prior to screening or who cannot stop using any tobacco products during the study.

  4. Subjects with a history of allergy to ≥ 2 drugs, or known hypersensitivity or intolerance to the IMP or similar products and their excipients.

  5. Presence of any suspected and/or definitively diagnosed malignancy at screening; or patients diagnosed with other malignancies within 5 years; 6. Previous or current medical history of cardiovascular, hematological, respiratory, digestive, urinary, endocrine/metabolic, neurological, or psychiatric disorders that, in the investigator's judgment, may affect the study outcomes.

  7. History of acute or chronic pancreatitis, biliary/gallbladder diseases , or pancreatic injury.

  8. Major surgery (including but not limited to procedures requiring general anesthesia) within 3 months prior to screening; or history of organ transplantation (except corneal transplantation performed more than 4 months prior to screening); or incomplete recovery from illness, trauma, or surgery at screening (e.g., significant impairment in daily living or working capacity compared to pre-illness/injury/surgery status); or planned surgery during the study period.

  9. Blood donation or significant blood loss (> 400 mL), or blood transfusion in the 3 months prior to screening.

  10. Presence of any clinically significant abnormalities in 12-lead electrocardiogram, vital signs (blood pressure, respiration, pulse rate, body temperature), physical examination, imaging examination, or laboratory tests (hematology, urinalysis, blood chemistry, coagulation function, serum amylase, serum lipase, calcitonin) as determined by the investigator at screening..

  11. Positive screening results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody infection at screening.

  12. History of organ transplantation, or acquired or congenital immune system disorders.

  13. Participation in a clinical study of another investigational medicinal product (IMP), surgery, or device within 3 months before screening, or within 5 half-lives of the previous IMP (whichever is longer). Or plan to participate in another clinical study of an IMP, surgery, or device before completing all scheduled assessments in the clinical study.

  14. Subjects who have used GLP-1 receptor agonists or drugs with the mechanism of action of GLP-1R agonists.

  15. Subjects who are allergic to any food or have specific dietary requirements and cannot adhere to a standardized diet.

  16. History of needle or blood phobia, or difficulty with blood collection; or inability/unwillingness to undergo repeated venipuncture.

  17. Subjects who were considered not suitable for the clinical study due to other reasons at the discretion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-08 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | Day 36 (end of period)
  Area under the plasma concentration-time curve at 0 h to last observation time-point after a single dose.

SECONDARY OUTCOMES:
AUC0-inf | Day 36 (end of period)
  Area under the plasma concentration-time curve at 0 h to infinity after a single dose.
TEAEs | Day 36 (end of period)
  Treatment-emergent adverse events in terms of number of subject
Hypoglycemia | Day 36 (end of period)
  Number of subjects, number of events and incidence of treatment-emergent hypoglycemia.
Immunogenicity | Day 36 (end of period)
  Including anti-drug antibody (ADA) and neutralizing antibody (NAb).
Cmax | Day 36 (end of period)
  Maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Study site 01, Beijing, China